CLINICAL TRIAL: NCT02182622
Title: Ib Dose Finding Study of LDE225 Plus Docetaxel/Prednisone in Patients With Advanced or Metastatic Castration Resistant Prostate Cancer Who Experience Disease Progression After Receiving Docetaxel
Brief Title: LDE225 + Docetaxel/Prednisone for Adv/Met Castrate Resistant Prostate Cancer w/ Disease Progression After Docetaxel
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Martin Gutierrez (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Martin Gutierrez, M.D., Director, Drug Discovery/Phase 1 unit, Hackensack Meridian Health
Organization: Hackensack Meridian Health (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-LDE225
Record Dates: First submitted 2014-06-27; First posted 2014-07-08 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level -1 (Experimental): Docetaxel 60mg/m2 IV every 21 days Prednisone 5mg oral twice daily LDE225 200mg oral daily
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: LDE225
- Dose Level 1 (Experimental): Docetaxel 75mg/m2 IV every 21 days Prednisone 5mg oral twice a day LDE225 200mg oral daily
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: LDE225
- Dose Level 2 (Experimental): Docetaxel 75mg/m2 IV every 21 days Prednisone 5mg oral twice daily LDE225 400mg oral daily
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: LDE225
- Dose Level 3 (Experimental): Docetaxel 75mg/m2 IV every 21 days Prednisone 5mg oral twice daily LDE225 800mg oral daily
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: LDE225

INTERVENTIONS:
Drug: Docetaxel
Drug: Prednisone
Drug: LDE225

SUMMARY:
The purpose of this study is to first determine the highest dose of LDE225 combined wtih Docetaxel and Prednisone that can be given that does not cause unacceptable side effects when given to patients with castrate resistant prostate cancer who failed previous docetaxel therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 18 years or older
* Histologically documented prostate adenocarcinoma with progressive systemic (clinically metastatic disease as documented in bone, CT or MRI scans) disease despite castrate levels of testosterone due to orchiectomy or Luteinizing-hormone-releasing hormone (LHRH) antagonist
* Must have received prior Docetaxel treatment with evidence of disease progression AND have at least one (e.g. Abiraterone Acetate, Enzalutamide, Cabazitaxel, Radium-223) of the four FDA approved therapies
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* At least one measurable site of disease (as defined by Response Evaluation Criteria in Solid Tumors) or other specific response assessment criteria as appropriate
* Able to swallow and retain oral medication
* Must have a castrate level of testosterone (=/< 50ng/dl or 1.7nmol/L). Castrate status must be maintained by continued gonadotropin-releasing hormone (GnRH) analogues unless patient has undergone surgical orchiectomy
* Discontinuation of all anti-androgen (except GnRH analogues - patients will continue on GnRH analogues to maintain castrate levels during study), anti-neoplastic or investigational treatment =/> 4 weeks (6 weeks for bicalutamide)
* Must have documented progressive disease to the previous line of therapy according to the Prostate Cancer Working Group 2 (PCWG2) criteria: patients who progressed based solely on Prostate Specific Antigen (PSA) rising, should have had a sequence of rising values on 3 consecutive occasions of at least 1 week intervals and should have 5.0ng/mL minimum level for entry; patients who manifested disease progression per the Response Evaluation Criteria in Solid Tumors (RECIST) are eligible independent of PSA; patients who manifest with bone only progressive disease, according to PCWG2 are eligible.
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9/L
* Hemoglobin (Hgb) ≥ 9 g/dL
* Platelets ≥ 80 x 10^9/L
* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Aspartate Aminotransferate (AST) and Alanine Transaminase (ALT) ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present
* Plasma creatine phosphokinase (CK) < 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50ml/min

Exclusion Criteria:

* Asymptomatic or minimally symptomatic patients with docetaxel naïve metastatic castration resistant prostate cancer
* Patients who have had major surgery within 4 weeks of initiation of study medication
* Patients with concurrent uncontrolled medical conditions that may interfere with their participation in the study or potentially affect the interpretation of the study data
* Patients unable to take oral drugs or with lack of physical integrity of the upper gastrointestinal tract or known malabsorption syndromes (e.g., ulcerative colitis, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patients who have previously been treated with systemic LDE225 or with other Hh pathway inhibitors
* Patients who have active uncontrolled or symptomatic central nervous system (CNS) metastases
* History of hypersensitivity to LDE225 or to drugs of similar chemical classes
* Patients who have neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as 3-hydroxy-3-methylglutaryl-coenzyme A (HMG CoA) inhibitors (statins), clofibrate and gemfibrozil, and that cannot be discontinued at least 2 weeks prior to starting LDE225 treatment. If it is essential that the patient stays on a statin to control hyperlipidemia, only pravastatin may be used with extra caution
* Patients who are planning on embarking on a new strenuous exercise regimen after initiation of study treatment: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on LDE225 treatment
* Patients who have taken part in an experimental drug study within 4 weeks or 5 half-lives, whichever is longer, of initiating treatment with LDE225
* Patients who are receiving other anti-neoplastic therapy besides Docetaxel (e.g. chemotherapy, targeted therapy or radiotherapy) concurrently or within 2 weeks of starting treatment with LDE225
* Patients who are receiving treatment with medications known to be moderate and strong inhibitors or inducers of Cytochrome P450 3A4/5 (CYP3A4/5) or drugs metabolized by Cytochrome P450 2B6 (CYP2B6) or Cytochrome P450 2C9 (CYP2C9) that have narrow therapeutic index, and that cannot be discontinued before starting treatment with LDE225. Medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A/5 inducers for at least 2 weeks prior to starting treatment with LDE225
* Patients who require the use of warfarin (substrate of CYP2C9) cannot be enrolled as LDE225 is a competitive inhibitor of CYP2C9 based on in-vitro data
* Impaired cardiac function or clinically significant heart disease, including any one of the following: Angina pectoris within 3 months Acute myocardial infarction within 3 months QTcF > 450 msec for males and > 470 msec for females on the screening ECG A past medical history of clinically significant ECG abnormalities or a family history of prolonged QT-interval syndrome Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Prior to study entry any ECG abnormality has to be documented by the investigator as not medically relevant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | From date of first dose until documentation of unacceptable toxicity or documented disease progression, whichever came first, assessed at up to days 42

CONTACTS AND LOCATIONS:
Locations (1):
- John Theurer Cancer @ HackensackUMC, Hackensack, New Jersey, United States